CLINICAL TRIAL: NCT02463253
Title: Correlation of Molecular Biomarkers With Biopsy Findings and Outcomes in Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: 665869
Record Dates: First submitted 2015-04-22; First posted 2015-06-04 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Delayed Graft Function
Keywords: Renal Biopsy; elevated serum creatinine; proteinuria
MeSH Terms: conditions — Delayed Graft Function; Proteinuria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Laboratory evaluations: The UC Davis laboratory will be used for clinical chemistry, and hematology, as well as other outside laboratories that the participants may go to
  1. Hematology: Routine hematological parameters will be analyzed as indicated by standard clinical care
  2. Clinical chemistry: Routine clinical chemistry parameters will be analyzed including basic and comprehensive metabolic profiles as indicated by standard clinical care Immunologic Profiles: As per standard routine monitoring with both indicated and surveillance biopsies, donor specific antibodies will be monitored
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Phase 1: A. OBJECTIVE: The objective of this phase of the study is to allow the clinical site to gain familiarity with patient recruitment, sample and data collection, and interpretation of the proteogenomic biomarker report provided, through retrospective analysis. This phase of the study will provide a platform for the transplant physicians to gain confidence with the format, logistics, and potential use of the biomarker tests on blood and tissue.
  B. STUDY DESIGN: Enroll 20 subjects who are post-transplant and are undergoing kidney transplant biopsies at the UC Davis transplant center. Ten subjects will be enrolled who are receiving surveillance "protocol biopsies" and 10 subjects.

SUMMARY:
This is a single-center, prospective, non-randomized, observational study to evaluate specific proteogenomic biomarker panels for acute rejection (AR) and chronic allograft nephropathy/interstitial fibrosis and tubular atrophy (CAN/IFTA) in blood, urine and kidney tissue (biopsy) in kidney transplant recipients. Proteogenomic profiles will be routinely monitored over one year after enrollment.

DETAILED DESCRIPTION:
OBJECTIVE: The objective of this phase of the study is to allow the clinical site to gain familiarity with patient recruitment, sample and data collection, and interpretation of the proteogenomic biomarker report provided, through retrospective analysis. This phase of the study will provide a platform for the transplant physicians to gain confidence with the format, logistics, and potential use of the biomarker tests on blood and tissue.

ELIGIBILITY:
Inclusion Criteria: Patients who meet all of the following criteria are eligible for enrollment as study participants:

1. Male and female recipients of all races, ≥18 years of age.
2. Patients undergoing primary or subsequent deceased-donor or living donor kidney transplantation.
3. Subject and/or guardian must be able to provide informed consent.
4. Subject and/or guardian must be able to comply with the study protocol.

Exclusion Criteria:

1. Need for combined organ transplantation with an extra-renal organ and/or islet cell transplant.
2. Recipients of previous non-renal solid organ and/or islet cell transplantation
3. Infection with HIV.
4. Inability or unwillingness of a participant and/or guardian to provide informed consent

   -

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: post-transplant and are undergoing kidney transplant biopsies at the UC Davis transplant center. Ten subjects will be enrolled who are receiving surveillance "protocol biopsies" and 10 subjects who will be receiving "for cause" biopsies in the setting of an elevated serum creatinine or proteinuria. Samples of blood, and formalin-fixed, paraffin-embedded biopsy tissue will be sent to Transplant Genomics INC. (TGI) for study purposes. In addition, clinical data will be collected on each subject.. Blood and tissue will be analyzed by TGI using Affymetrix microarrays, and reports will be sent to UC Davis retrospectively. Samples may be batch-shipped and results will not be reported in real time. These results will be compared to both the histological diagnosis, and to the clinical course.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Biopsy prove acute rejection | 12 months
  Incidence of acute rejection at the time of any kidney biopsy

SECONDARY OUTCOMES:
Gene Expression Profiling | 12 months
  Blood and tissue collection from each subject at the time of each for cause or protocol kidney biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Angelo DeMattos, MD, Principal Investigator — University of California, Davis Health Systems
Locations (1):
- University of California, Davis Transplant Center, Sacramento, California, United States